CLINICAL TRIAL: NCT03483259
Title: To Explore the Pharmacokinetics and Relative Bioavailability of Sulfatinib Capsules in Two Different Manufacturers in Chinese Adult Male Healthy Volunteers
Brief Title: To Explore the Pharmacokinetics and Relative Bioavailability of Sulfatinib Capsules in Two Different Manufacturers
Acronym: CRC-C1721
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-012-00CH2
Record Dates: First submitted 2018-03-08; First posted 2018-03-30 (Actual); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Relative Bioavailability
Keywords: Pharmacokinetics; Relative bioavailability
MeSH Terms: interventions — surufatinib

STUDY DESIGN:
Intervention Model Description: Eligible subjects who did not meet the exclusion criteria were randomly assigned to one of the three groups: group A, B, and C (administration TRR, RTR and RRT, 9 subjects in each group, where T is the test formulation and R is the reference formulation) .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A-Sulfatinib T capsule (Experimental): The subjects in this arm will receive sulfatinib T capsules from Hutchison Whampoa Pharmaceutical (Suzhou) Co., Ltd.
  Interventions: Drug: Sulfatinib T capsule
- Arm B-Sulfatinib R capsule (Experimental): The subjects in this arm will receive sulfatinib R capsules from Beijing Yiling Bioengineering Technology Co., Ltd.
  Interventions: Drug: Sulfatinib R capsule

INTERVENTIONS:
Drug: Sulfatinib T capsule — Sulfatinib T capsules were produced by Hutchison Whampoa Pharmaceutical (Suzhou) Co., Ltd. production.
  Other Names: HMPL-012, Surufatinib
  Arms: Arm A-Sulfatinib T capsule
Drug: Sulfatinib R capsule — Sulfatinib R capsules were produced by Beijing Yiling Bioengineering Technology Co., Ltd.
  Other Names: HMPL-012, Surufatinib
  Arms: Arm B-Sulfatinib R capsule

SUMMARY:
This is a single-center, randomized, open, single-dose, three-cycle cross-design study, which will be only enrolled Chinese male healthy volunteers.

DETAILED DESCRIPTION:
27-30 Chinese male healthy volunteers will be enrolled to assess the pharmacokinetic profile and relative bioavailability of 300 mg (50 mg x 6) Sulfatinib capsules of single dose orally in two different manufacturers after breakfast. All subjects are required to collect PK blood samples before and after administration at the following time points: within 1 hour before administration, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 12, 24, 36, 48, 72, 96 hours after administration (16 times point), each collection of venous blood is 2mL.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be voluntary and sign an informed consent form and agree to comply with the requirements of the protocol；
2. Age of 18-40 (inclusive), male healthy volunteers；
3. Medical history, physical examination, 12-lead ECG and laboratory tests at screening judged as normal or abnormal but not clinically significant by investigators;
4. Medical history, physical examination, 12-lead ECG and laboratory tests at screening judged as normal or abnormal but not clinically significant by investigators;
5. Men whose partners are women of childbearing potential are required to use adequate contraceptive methods during participation in this study；

Exclusion Criteria:

1. Any clinically significant disease or condition includes but not limited to metabolism/endocrine, liver, kidney, blood, lung, immune, cardiovascular, gastrointestinal, genito-urinary, nervous, or mental illness that judged by the investigator within 3 months before screening;
2. Previous gastrointestinal surgery, kidney surgery, cholecystectomy and surgery history may affect the absorption or excretion of drugs;
3. Hypertension: systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg;
4. Hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV Ab) test positive, HIV or treponema pallidum antibodies test positive;
5. Any drugs that may change the liver and kidney clearance;
6. Take any prescription drug (including Chinese herbal medicine) within 14 days before dosing; or use any over-the-counter drugs (including but not limited to vitamins, prophylaxis, plant health products) within 7 days before dosing;
7. Clinical trials of other medications before screening, less than a 5-fold half-life or 28 days from the time of the last other study drug, whichever is longer;
8. Any history of clinically serious disease or condition that the investigator believes may affect the outcome of this study.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2018-05-12 (Actual); Study Completion 2018-05-18 (Actual)

PRIMARY OUTCOMES:
The area under the plasma concentration-time curve (AUC) from 0 to the time of the last measurable concentration (AUCt) of Sulfatinib | Measured on the Cycle1 Day1 to Day5, Cycle2 Day1 to Day5, Cycle3 Day1 to Day5
  The area under the plasma concentration-time curve (AUC) from 0 to the time of the last measurable concentration.
Maximum observed plasma concentration (Cmax) of Sulfatinib | Measured on the Cycle1 Day1 to Day5, Cycle2 Day1 to Day5, Cycle3 Day1 to Day5
  Maximum observed concentration, occurring at Tmax.
The time to Cmax (peak time, Tmax) of Sulfatinib | Measured on the Cycle1 Day1 to Day5, Cycle2 Day1 to Day5, Cycle3 Day1 to Day5
  The time at which maximum plasma concentration (Cmax) is observed.
Half-life (t1/2) of Sulfatinib | Measured on the Cycle1 Day1 to Day5, Cycle2 Day1 to Day5, Cycle3 Day1 to Day5
  The time required for the concentration of the drug to reach half of its original value.
Relative Bioavailability | Measured on the Cycle1 Day1 to Day5, Cycle2 Day1 to Day5, Cycle3 Day1 to Day5
  This term represents the relationship between the bioavailability of a substance in two different media.

SECONDARY OUTCOMES:
Adverse Event (AE) monitoring of Sulfatinib | Measured from the date signed ICF to within 14 days after the last dose
  AE monitoring will be assessed by incidence of AEs, AE grading, serious AEs, as well as laboratory determinations and vital sign parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Liu Yanmei, Master, Principal Investigator — Shanghai Xuhui District Central Hospital
Locations (1):
- Shanghai Xuhui District Central Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No